CLINICAL TRIAL: NCT05720286
Title: Verification of the Performance and Safety of the First Row Resorbable Threaded Anchor FIXIT® in Arthroscopic Rotator Cuff Repair as Part of the Post-marketing Follow-up of Device
Brief Title: Performance and Safety of the FIXIT® Anchor in Arthroscopic Rotator Cuff Repair
Acronym: FIXIT®2018
Status: Completed | Type: Observational
Sponsor: Science and biomaterials (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-A02653-52
Record Dates: First submitted 2023-01-27; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study group: There was only one group as the study was a non-comparative study
  Interventions: Device: Arthroscopic rotator cuff repair

INTERVENTIONS:
Device: Arthroscopic rotator cuff repair — Arthroscopic transosseous reinsertion of the rotator cuff is the most widely used arthroscopic technique. The tendons are repositioned on the greater and lesser tuberosities of the humerus with specific anchors. These anchors, placed in the humeral bone, are attached to sutures which are in turn tied to the tendon.

SUMMARY:
Verification of the performance and safety of the first row resorbable threaded anchor FIXIT® in arthroscopic rotator cuff repair Non-interventional, prospective, non-comparative, multi-center study as part of the post-marketing follow-up of devices

DETAILED DESCRIPTION:
the main objective of this study was to verify the safety of the resorbable threaded anchor FIXIT®, used in arthroscopic rotator cuff repair. This objective was to be imaging assessed (echography, MRI) for the presence or absence of a rotator cuff re-tear and its degree of retractation. The second objective was to verify the performance of the FIXIT® anchor with 4 scoring criteria : Constant score, pain score EVA, Quick DASH score and Bernageau classification

ELIGIBILITY:
Inclusion Criteria:

* Patient with broken tendinopathy of the rotator cuff
* Patient over 18 years old
* Patient who has received complete medical information and not objecting to participate in research
* Social insured patient

Exclusion Criteria:

* Pregnant or likely to be pregnant, or breastfeeding
* Patient under guardianship
* Non-cooperative patient, who does not want or is unable to follow the post-operative instructions (drug addict or alcoholic patient in particular)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 patients, aged between 45 to 78 and operated for a rotator cuff repair were selected in this study. Initially, 31 patients were included but 1 withdrew from the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Sugaya classification | 1 year postoperative
  Radiological evaluation to assess the absence of rotator cuff re-tears with the Sugaya classification and the retraction's degree of the cuff.

SECONDARY OUTCOMES:
Constant score | 45 days, 5months and 1 year postoperative
  Functional score
Pain score | 45 days, 5months and 1 year postoperative
  EVA pain scale
Quick DASH score | 45 days, 5months and 1 year postoperative
  Capacity of shoulder score
Fatty degeneration | preoperative
  Bernageau classification

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BONNEVIALLE, Pr, Principal Investigator
Locations (2):
- France (2):
  - Polyclinique de l'Ormeau, Tarbes
  - CH Purpan, Toulouse